CLINICAL TRIAL: NCT02755623
Title: Structural and Functional Correlates of Clinical Response to Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment in Schizophrenia Patients With Resistant Auditory Hallucinations
Brief Title: Structural and Functional Correlates of Clinical Response to rTMS Treatment in Schizophrenia Patients With Resistant Auditory Hallucinations
Acronym: TMSCCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Dominique JANUEL, head of research center and clinical professor, Centre hospitalier de Ville-Evrard, France
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dmdpt6tech/mm/2014-A01595-42
Record Dates: First submitted 2016-04-22; First posted 2016-04-29 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Repetitive Transcranial Magnetic Stimulation (rTMS) (Active Comparator): low-frequency (1 Hertz) rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham Repetitive Transcranial Magnetic Stimulation (rTMS) (Sham Comparator): sham TMS
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Participants are sequentially randomly assigned to either 20 active rTMS sessions or 20 sham rTMS sessions that were applied over the left temporoparietal junction. Treatments are administered daily, over a period of two weeks.
  Arms: Active Repetitive Transcranial Magnetic Stimulation (rTMS)
Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)
  Arms: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)

SUMMARY:
The potential of non-invasive Transcranial Magnetic Stimulation (TMS) as a therapeutic tool for improving schizophrenic symptoms, in particular resistant hallucinations, has been increasingly studied over the past decades. Several studies have demonstrated that low-frequency patterns of repetitive TMS (rTMS) applied over the left Temporoparietal Junction (TPJ), which are known to decrease local activity, significantly reduced auditory verbal hallucinations in schizophrenic patients. In spite of highly promising results, a high level of inter-individual variability in the responses to non-invasive brain stimulation treatments, and the fact that rTMS may prove ineffective in some patients, keep spurring controversy about the efficacy of these approaches (as currently performed), as well as about how to increase its efficacy and consistency. Accordingly, the objectives of this project are to better understand the impact of rTMS on the brains of patients with resistant auditory hallucinations, and to use this information not only to better understand this condition but to develop more efficient and consistent therapies. Thus, in this study, the investigators focus more specifically on resistant auditory hallucinations in schizophrenia, which is a common symptom in schizophrenic patients, and can be treated by rTMS. The investigators hypothesize that there is a baseline difference in anatomical and/or functional connectivity between responder and non-responder patients who are treated with rTMS. Therefore, our project will aim to determine some anatomical and functional connectivity markers of response to rTMS treatment in patients with schizophrenia

DETAILED DESCRIPTION:
The potential of non-invasive Transcranial Magnetic Stimulation (TMS) as a therapeutic tool for improving schizophrenic symptoms, in particular resistant hallucinations, has been increasingly studied over the past decades. Several studies have demonstrated that low-frequency patterns of repetitive TMS (rTMS) on the left temporoparietal junction (TPJ), which are known to decrease local activity, significantly reduce auditory verbal hallucinations in schizophrenic patients. In spite of highly promising results, a high level of inter-individual variability in the response to non-invasive brain stimulation treatments, and the fact that rTMS may prove ineffective in some patients, keep spurring controversy on the efficacy of these approaches as currently performed, and on how to increase its efficacy and consistency. To date, few studies have aimed to explain this variability when, in fact, a better understanding of this common phenomena in the neurostimulation domain would clearly increase the effectiveness of this treatment, and lead to individualized therapeutic approaches specifically tailored to the conditions of each patient. Moreover, many questions stand, particularly regarding the influence of rTMS treatment on the anatomical and functional connectivity in schizophrenic patients.

Accordingly, the objectives of this project are to better understand the impact of rTMS on the brains of patients with resistant auditory hallucinations, and to use this information not only to better understand this condition but to develop more efficient and consistent therapies. The investigators hypothesize that there is a baseline difference in anatomical and/or functional connectivity between responder and non-responder patients who are treated with rTMS. Therefore, this project aims to determine some anatomical and functional connectivity markers of response to rTMS treatment in patients with schizophrenia. For this, the investigators compare the patterns of diffusion tensor imaging (DTI) white matter tractography and resting-state functional magnetic resonance imaging (fMRI) data between responder and non-responder patients to rTMS treatment. Moreover, the investigators believe that rTMS can increase the functional connectivity between frontal and temporo-parietal cortices in schizophrenic patients associated with improvements in auditory hallucinations. Therefore, the second objectives of this work are to evaluate the impact of rTMS in functional connectivity in patients with schizophrenia by comparing the DTI and resting-state fMRI data before and after rTMS treatment in both responder and non-responder patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of schizophrenia according to DSM-V (Diagnostic and Statistical Manual of Mental Disorder V, 2013) criteria
* Clinically stabilized for at least 3 months
* Patient with resistant auditory hallucinations
* Male or female, 18 to 65 years old
* A written agreement from the patient's legal guardian/s, if applicable
* Right-handed
* A good knowledge of the French language
* Signed consent form

Exclusion Criteria:

* Other diseases than schizophrenia
* Indulging in an addiction (alcohol, psychoactive substances) over the last 12 months
* Patient who has received rTMS treatment in the last 12 months
* Patient who is participating in a concurrent research protocol
* Patient with a history of seizures
* rTMS contraindications: patient with epilepsy, brain surgery and/or head trauma in the past, use of cardiac pacemaker, or surgical staples on the scalp
* MRI contraindications: pregnancy or lactating (n.b. a negative pregnancy test will be required if the patient is a female in reproductive years who does not use contraception); use of cardiac pace maker or surgical staples; patient with a neurological disorder, head trauma or claustrophobia
* Patient with severe cardiovascular disease
* Patient with medication which reduces the epileptic threshold (bupropion, methadone and theophylline)
* Patients placed in psychiatric care either by the state or a third party

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-10-14 (Actual); Primary Completion 2025-09-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Changes in the integrity of white matter tracts between responder and non-responder patients | Baseline
Changes in the variations of the blood-oxygen-dependent level (BOLD) signal between responder and non-responder patients | Baseline

SECONDARY OUTCOMES:
AHRS (Auditory Hallucinations Rating Scale) | Baseline, 3 weeks, 7 weeks and 15 weeks
HCS (Hallucinations Change Score) | Baseline, 3 weeks, 7 weeks and 15 weeks
PANSS (Positive And Negative Syndrome Scale) | Baseline, 3 weeks, 7 weeks and 15 weeks
PSYRATS (Psychotic Symptom Rating Scale) | Baseline, 3 weeks, 7 weeks and 15 weeks
BDI (Beck Depression Inventory) | Baseline, 3 weeks, 7 weeks and 15 weeks
Serum BDNF levels | Baseline, 3 weeks, 7 weeks and 15 weeks
Measure of the amplitude of Motor-Evoked Potentials (MEPs) | Baseline, 3 weeks, 7 weeks and 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Thomas, BIOLOGISTE, Principal Investigator — Unité de Recherche Clinique, EPS Ville Evrard, Neuilly-sur-Marne,, France, 93330; Dominique Januel, MD, PhD, Principal Investigator — Unité de Recherche Clinique, EPS Ville Evrard, Neuilly-sur-Marne,, France, 93330
Locations (1):
- Unité de Recherche Clinique, EPS Ville Evrard, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas F, Bouaziz N, Gallea C, Schenin-King Andrianisaina P, Durand F, Bollore O, Benadhira R, Isaac C, Braha-Zeitoun S, Moulier V, Valero-Cabre A, Januel D. Structural and functional brain biomarkers of clinical response to rTMS of medication-resistant auditory hallucinations in schizophrenia patients: study protocol for a randomized sham-controlled double-blind clinical trial. Trials. 2019 Apr 23;20(1):229. doi: 10.1186/s13063-019-3311-x. PMID 31014369